CLINICAL TRIAL: NCT07351942
Title: Clinical and Ultrasonographic Evaluation of the Effectiveness of Low-Load Resistance Training With Blood Flow Restriction in the Treatment of Lateral Epicondylitis: A Randomized, Double-Blind, Controlled Trial
Brief Title: Effectiveness of Low-Load Resistance Training With Blood Flow Restriction in Lateral Epicondylitis
Acronym: LE-LLRT-BFR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Süleyman Çağlar Tekin, MD, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LE-LLRT-BFR-TR-34-SE-01
Record Dates: First submitted 2026-01-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; Tennis Elbow; Blood Flow Restriction Training; BFR; Low-Load Resistance Training; Exercise Therapy; Ultrasonography
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups and receive the same low-load resistance exercise program either with a blood flow restriction procedure or with a sham blood flow restriction procedure throughout the study period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are blinded to group allocation. Exercise sessions are supervised by therapists who are not involved in outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Load Resistance Training with Blood Flow Restriction (Experimental): Participants receive a low-load resistance exercise program performed with a blood flow restriction procedure.
  Interventions: Other: Low-Load Resistance Training with Blood Flow Restriction
- Low-Load Resistance Training with Sham Blood Flow Restriction (Active Comparator): Participants receive the same low-load resistance exercise program performed with a sham blood flow restriction procedure.
  Interventions: Other: Low-Load Resistance Training with Sham Blood Flow Restriction

INTERVENTIONS:
Other: Low-Load Resistance Training with Blood Flow Restriction — A supervised low-load resistance training program performed with a blood flow restriction procedure applied to the affected upper extremity.
  Other Names: BFR Training
  Arms: Low-Load Resistance Training with Blood Flow Restriction
Other: Low-Load Resistance Training with Sham Blood Flow Restriction — A supervised low-load resistance training program performed with a sham blood flow restriction procedure applied to the affected upper extremity.
  Arms: Low-Load Resistance Training with Sham Blood Flow Restriction

SUMMARY:
Lateral epicondylitis, commonly known as tennis elbow, is a frequent musculoskeletal condition that causes pain, reduced grip strength, and functional limitations in daily activities. Exercise-based rehabilitation is a key component of treatment; however, the optimal exercise approach remains uncertain. Low-load resistance training combined with blood flow restriction (LLRT-BFR) has emerged as a promising method that may enhance training effects while using lower exercise loads, potentially reducing mechanical stress on the affected tissues while providing benefits comparable to high-load resistance training.

The purpose of this study is to evaluate the clinical and ultrasonographic effects of LLRT-BFR in patients with lateral epicondylitis. Adults aged 18-65 years with a recent diagnosis of lateral epicondylitis who meet predefined inclusion and exclusion criteria will be enrolled and randomly assigned to one of two exercise-based treatment groups. Both groups will participate in the same supervised low-load resistance exercise program, while one group will perform the exercises with blood flow restriction and the other group will receive a sham application without meaningful blood flow restriction.

Participants will undergo supervised exercise sessions twice weekly for six weeks. Outcomes will be assessed at baseline, on the first day after completion of treatment, and at 4 and 12 weeks during follow-up. The primary outcome will focus on functional status, while secondary outcomes will include pain intensity, pain sensitivity, grip strength, ultrasonographic measurements of tendon and muscle structure, and patient-reported treatment satisfaction.

By comparing these two exercise approaches, this study aims to provide evidence regarding the effectiveness and safety of LLRT-BFR and to clarify its potential role in the rehabilitation of patients with lateral epicondylitis.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of low-load resistance training with blood flow restriction (LLRT-BFR) in patients with lateral epicondylitis using clinical and ultrasonographic assessments.

Patients aged 18-65 years who present to the Physical Medicine and Rehabilitation outpatient clinic at Sisli Hamidiye Etfal Training and Research Hospital with elbow pain lasting longer than 2 weeks and shorter than 12 weeks will be screened for eligibility. A clinical diagnosis of lateral epicondylitis will be established by a physician based on localized pain at the tenoperiosteal junction of the common extensor tendon (CET) at the lateral epicondyle (LE) and its surrounding area, tenderness on palpation, pain elicited by provocation tests, including resisted wrist extension and resisted third finger extension, reduced grip strength, and impairment in activities of daily living. Patients who meet the inclusion criteria and provide informed consent will be enrolled.

Eligible participants will be randomly allocated into two groups using a computerized randomization program, with stratification based on sex, age, and upper extremity dominance. These two groups will be an experimental group receiving low-load resistance training with blood flow restriction (LLRT-BFR) and a control group receiving the same low-load resistance training with sham blood flow restriction (LLRT-Sham BFR).

In the LLRT-BFR treatment group, individualized arterial occlusion pressure (AOP) will be determined prior to each session. A pneumatic cuff will be placed at the most proximal region of the upper extremity, just distal to the deltoid muscle insertion. During exercise, cuff pressure will be set at a standardized level corresponding to 40% of the measured AOP, in accordance with previously published protocols. Participants in this group will undergo supervised LLRT-BFR sessions twice weekly for 6 weeks, totaling 12 sessions.

In the LLRT-Sham BFR control group, individualized arterial occlusion pressure (AOP) will also be determined prior to each session. A pneumatic cuff will be placed at the most proximal region of the upper extremity, just distal to the deltoid muscle insertion, in the same manner as in the experimental group. During exercise, the cuff will be applied without intentional inflation; any pressure present will be limited to that resulting from cuff placement alone and will be substantially lower than the individually determined arterial occlusion pressure (AOP), and insufficient to induce meaningful blood flow restriction. Participants in this group will undergo supervised LLRT-Sham BFR sessions twice weekly for 6 weeks, totaling 12 sessions.

AOP will be assessed while the patient is seated comfortably, using a pneumatic cuff and Doppler ultrasonography with a linear ultrasound probe suitable for musculoskeletal examination to detect radial artery pulsation. Care will be taken to apply minimal probe pressure to avoid influencing AOP measurements. The cuff pressure at which Doppler activity due to radial artery pulsation is no longer detectable will be recorded as the AOP. During exercise, cuff pressure will be applied according to group allocation and maintained throughout each exercise set, and released between different exercises, allowing continued arterial inflow while temporarily restricting venous outflow in a controlled and safe manner.

Each treatment session will include approximately 45 minutes of supervised exercise therapy conducted in accordance with routine clinical practice. The exercise program will consist of low-load strengthening exercises for wrist flexion and extension, forearm pronation and supination, and wrist radial and ulnar deviation, as well as stretching exercises targeting the wrist flexor and extensor muscle groups. Exercises will be performed in a 3x10 repetition scheme, with 30-second rest intervals between sets and 90-second rest intervals between exercises targeting different muscle groups.

Clinical and ultrasonographic assessments will be conducted at baseline (pre-treatment), on the first day after treatment completion, and at 4 and 12 weeks post-treatment. The primary outcome measure will be functional status assessed using the Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire. Secondary outcome measures will include pain intensity assessed by visual analog scale (VAS) during movement, at rest, at night, and during maximal grip; pain sensitivity assessed as pressure pain threshold using an algometer; maximal and pain-free grip strength assessed using a handheld dynamometer; ultrasonographic measurements of common extensor tendon thickness obtained at standardized anatomical locations (1 cm distal to the lateral epicondyle, capitellar region, and radiocapitellar region); cross-sectional area measurements of the extensor carpi radialis brevis and extensor digitorum communis muscles performed at a standardized level corresponding to 40% of the forearm length measured distally from the lateral epicondyle toward the Lister tubercle; the Total Ultrasonography Scale Score evaluating predefined tendon characteristics (e.g., hypoechogenicity, neovascularization, heterogeneity, and bony abnormalities); and treatment satisfaction assessed using the Roles-Maudsley Score.

The influence of demographic and anthropometric variables, including sex, age, height, weight, body mass index (BMI), and upper extremity dominance, on outcome measures will also be analyzed.

Randomization will be performed using a computerized randomization program by a non-evaluating research assistant who will be aware of group allocation and responsible for data recording. Blinding will be ensured by keeping participants unaware of their group assignment and by maintaining outcome assessors blinded to group allocation throughout the study. The study is designed as a single-center, prospective, randomized, double-blind, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of lateral epicondylitis established by a physician
* Presence of symptoms consistent with lateral epicondylitis for more than 2 weeks and less than 12 weeks
* Adults aged 18 to 65 years
* Visual Analog Scale (VAS) pain score ≥ 3
* Willingness to participate in the study and provision of written informed consent

Exclusion Criteria:

* History of major trauma to the elbow or surrounding region within the past 1 month
* Receipt of physical therapy for the elbow or surrounding region within the past 1 year
* History of corticosteroid or other injection therapies to the elbow or surrounding region within the past 1 year
* History of fracture involving the elbow or surrounding region
* History of surgery involving the elbow or surrounding region
* Presence of rheumatologic diseases affecting the elbow or surrounding region
* History of peripheral vascular disease
* History of coagulation disorders
* History of severe cardiovascular disease
* History of uncontrolled hypertension
* History of uncontrolled diabetes mellitus
* Clinical findings consistent with cervical radiculopathy causing elbow pain or muscle weakness in the affected upper extremity
* Clinical findings consistent with shoulder pathologies causing elbow pain or muscle weakness in the affected upper extremity
* Restricted range of motion of the elbow joint detected on clinical examination
* History of severe psychiatric disorders
* History of malignancy
* Pregnancy
* Unwillingness to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation (PRTEE) Total Score | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire is used to assess pain and functional disability related to lateral epicondylitis. The total score ranges from 0 to 100, with higher scores indicating greater pain and functional impairment.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Pain Intensity Scores | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  Pain intensity assessed using a Visual Analog Scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain, with higher scores representing greater pain intensity, for pain during activity, at rest, at night, and during maximal grip.
Pressure Pain Threshold | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  Pressure pain threshold is assessed using an algometer applied over the lateral epicondyle region to evaluate pain sensitivity.
Grip Strength | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  Maximal grip strength and pain-free grip strength are measured using a handheld dynamometer to assess functional hand strength.
Common Extensor Tendon Thickness | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  Ultrasonographic measurement of common extensor tendon thickness performed at three standardized locations: 1 cm distal to the lateral epicondyle, the capitellar region, and the midpoint of the radiocapitellar joint line.
Cross-Sectional Area of the Extensor Carpi Radialis Brevis and Extensor Digitorum Communis Muscles | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  Ultrasonographic measurement of the cross-sectional area of the extensor carpi radialis brevis and extensor digitorum communis muscles performed at a standardized level corresponding to 40% of the forearm length, measured distally from the lateral epicondyle toward the Lister tubercle. Measurements are performed separately for each muscle.
Total Ultrasonography Scale Score (TUSS) | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  Structural changes of the common extensor tendon assessed using the Total Ultrasonography Scale Score (TUSS), a composite ultrasonographic score ranging from 0 to 8, based on predefined tendon characteristics including hypoechogenicity (0-3), neovascularization (0-3), heterogeneity (0-1), and bony abnormalities (0-1). Higher scores represent greater structural tendon pathology.
Roles-Maudsley Score (RMS) | Baseline (pre-treatment), Day 1 post-treatment, Week 4 post-treatment, and Week 12 post-treatment
  Pain and functional limitation during daily activities assessed using the Roles-Maudsley Score (RMS), a four-point ordinal scale based on patient self-assessment, ranging from 1 to 4, where 1 indicates excellent function with no pain and 4 indicates poor function with severe pain, with higher scores representing greater pain and functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Çağlar Tekin, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as this is a single-center, academic study, and there is no plan or requirement to make the raw dataset publicly available.

REFERENCES:
- [Background] Krogh TP, Fredberg U, Ammitzboll C, Ellingsen T. Clinical Value of Ultrasonographic Assessment in Lateral Epicondylitis Versus Asymptomatic Healthy Controls. Am J Sports Med. 2020 Jul;48(8):1873-1883. doi: 10.1177/0363546520921949. Epub 2020 Jun 2. PMID 32484714
- [Background] Toprak U, Baskan B, Ustuner E, Oten E, Altin L, Karademir MA, Bodur H. Common extensor tendon thickness measurements at the radiocapitellar region in diagnosis of lateral elbow tendinopathy. Diagn Interv Radiol. 2012 Nov-Dec;18(6):566-70. doi: 10.4261/1305-3825.DIR.5575-12.2. Epub 2012 Apr 13. PMID 22498913
- [Background] Bechan Vergara I, Puig-Divi A, Amestoy Alonso B, Mila-Villarroel R. Effects of low-load blood flow restriction training in healthy adult tendons: A systematic review and meta-analysis. J Bodyw Mov Ther. 2024 Jul;39:13-23. doi: 10.1016/j.jbmt.2023.11.048. Epub 2023 Dec 3. PMID 38876617
- [Background] Karanasios S, Korakakis V, Moutzouri M, Xergia SA, Tsepis E, Gioftsos G. Low-Load Resistance Training With Blood Flow Restriction Is Effective for Managing Lateral Elbow Tendinopathy: A Randomized, Sham-Controlled Trial. J Orthop Sports Phys Ther. 2022 Dec;52(12):803-825. doi: 10.2519/jospt.2022.11211. Epub 2022 Sep 13. PMID 36099170